CLINICAL TRIAL: NCT06733922
Title: Exploratory Evaluation of Novel Investigational Eye Movement Biomarkers to Track Ofatumumab Treatment Response in Canadian Patients With Active Relapsing-Remitting Multiple Sclerosis (ELIOS)
Brief Title: ELIOS - Investigational Biomarkers to Track Disease Modification in Active RRMS
Acronym: ELIOS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COMB157GCA05
Record Dates: First submitted 2024-11-12; First posted 2024-12-13 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
Keywords: Ofatumumab; Eye Movement Biomarkers (EMB); Patient-Reported Outcomes (PRO); Active Relapsing-Remitting MS (RRMS); Real-World, Neurofilament Light Chain (NfL); Digital, Eye-Tracking
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Intervention Model Description: This is a Phase IV, interventional, multi-center, single-arm, open-label, exploratory, descriptive study conducted across geographical regions of Canada to assess the value of novel investigational Eye Movement Biomarkers (EMBs) in tracking disease-related changes among a real-world cohort of Canadian patients with active RRMS initiating ofatumumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETNATM-ProgMS (Experimental): Patients with active RRMS being prescribed ofatumumab as part of routine clinical care will have their eye movements reliably and accurately tracked using ETNATM-ProgMS SaMD (v1.0.11 or later) at baseline, 3-, 6-, 12-, and 24-months following ofatumumab initiation
  Interventions: Device: ETNATM-ProgMS

INTERVENTIONS:
Device: ETNATM-ProgMS — To that end, the study will use the patented investigational ETNATM-ProgMS SaMD (v1.0.11 or later), which has not yet received Health Canada approval, to reliably and accurately track eye movements with precision. Of note, investigational versions of this SaMD are used for the purpose of clinical research only and will not be commercialized.

SUMMARY:
The exploratory ELIOS study aims to assess the value of novel investigational Eye Movement Biomarkers (EMBs) in tracking disease-related changes among a real-world cohort of Canadian patients with active RRMS, within the context of disease-modifying treatment (i.e., ofatumumab). To that end, the study will use the patented investigational, Eye Tracking Neurological Assessment (ETNA-ProgMS) SaMD (v1.0.11 or later), which has not yet received Health Canada approval, to reliably and accurately track eye movements with precision.

ELIGIBILITY:
Inclusion criteria

Patients eligible for inclusion in the study must fulfill all of the following criteria:

1. Adult patients who are prescribed ofatumumab as part of routine clinical care as per the PM but who have not yet received their first dose. The decision to prescribe ofatumumab must be made prior to and independent of study participation.
2. Patients or their legally authorized representatives who sign the Institutional Review Boards/Independent Ethics Committee (IRB/IEC)-approved informed consent form.
3. Patients who meet the EDSS score range of 0 up to 7 at the time of screening and enrollment for ofatumumab treatment.
4. Patients with a diagnosis of active RRMS according to the 2017 Revised McDonald criteria2.
5. Patients who can provide blood samples.
6. Patients who can understand written and spoken Canadian English or French.
7. Patients who have sufficient corrected visual acuity to allow for accurate reading of the on-screen visual task instructions, in the judgement of the Investigator. If a relapse temporarily affects a patient's corrected visual acuity, the Baseline Visit may be postponed until the patient can accurately read the on-screen visual task instructions, if deemed acceptable by the Investigator and the patient.
8. Patients with a confirmed diagnosis of MS with no signs of progressive increase in physical disability independent of relapse activity within the past six months, as assessed by a physician.

Exclusion criteria

In order to ensure that the study population will be representative of all eligible patients, no additional exclusions may be applied by the Investigator. Patients meeting any of the following criteria are not eligible for inclusion in this study:

1. Patients with primary progressive MS, secondary progressive MS without disease activity, clinically isolated syndrome, or radiologically isolated syndrome.
2. Any disease or condition that could interfere with participation in the study according to the study protocol, or with the ability of the patients to cooperate and comply with the study procedures.
3. Pregnant or nursing (lactating) women.
4. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception while taking ofatumumab and for six months after stopping medication. Effective contraception methods include:

   * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
   * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks prior to enrollment. In case of oophorectomy alone, the reproductive status of the woman must be confirmed by follow-up hormone level assessment
   * Male sterilization at least six months prior to enrollment. For female participants on the study, the vasectomized male partner should be the sole partner for that participant
   * Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception, placement of an intrauterine device or intrauterine system, or other forms of hormonal contraception that have comparable efficacy (failure rate <1%) such as hormone vaginal ring or transdermal hormone contraception
   * Use of barrier methods of contraception (male or female condom, occlusive cap, diaphragm or cervical/vault caps)
   * In case of use of hormonal contraception women participants should have been stable on the same method for a minimum of three months before taking study treatment.
   * If local regulations are more stringent than the contraception methods listed above, local regulations apply and will be described in the ICF.
   * Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age-appropriate history of vasomotor symptoms). Women participants are considered not of child-bearing potential if they are post-menopausal or have had bilateral tubal ligation, surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral salpingectomy at least six weeks prior to first dose of study treatment on study. In the case of oophorectomy alone, a woman is not considered to be of child-bearing potential only when the reproductive status has been confirmed by follow-up hormone level assessment.
5. Patients with hypersensitivity to ofatumumab or to any ingredient in the formulation, active hepatitis B virus, progressive multifocal leukoencephalopathy (PML), severe active infections, in a severely immunocompromised state or with known active malignancies.
6. Patients with an active chronic disease (or stable but treated with immune therapy) of the immune system other than MS (e.g., rheumatoid arthritis, scleroderma, Sjögren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with immunodeficiency syndrome (hereditary immune deficiency, drug-induced immune deficiency).
7. Patients who are using other investigational drugs within 30 days prior to or at the Baseline Visit, or within a period corresponding to five elimination half-lives, whichever is longer, or who are using other investigational drugs for which the expected pharmacodynamic effect has not returned to baseline.
8. Contraindication or inability to undergo regular testing (e.g., MRI, blood tests) as per standard of care.
9. Patients who have been treated with cladribine or with alemtuzumab at any time within the 12 months prior to the Baseline Visit.
10. Patients who have had any prior exposure to anti-CD20 B-cell therapy (i.e., ocrelizumab, ofatumumab) or natalizumab.
11. Medical history or evidence of health issues that, in the opinion of the Investigator, may affect movements and oculomotor control.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
1- Change Eye Movement Biomarkers (EMB) | 6 months from baseline
  Change in subtle eye movement anomalies referred to as Eye Movement Biomarkers (EMBs). EMB are derived from composite scores of various Eye Movement metrics. Results stratified by patients experiencing a clinically meaningful change (CMC) in at least one traditional MS outcome (CMCp) or no CMC in all traditional MS outcomes (CMCs/i) at 24 months (or at the time of ofatumumab discontinuation and treated with ofatumumab for at least 12 months)

SECONDARY OUTCOMES:
1a. Change in EMB | 3,12 and 24 months from Baseline
  Change in subtle eye movement anomalies referred to as Eye Movement Biomarkers (EMBs). EMB are derived from composite scores of various Eye Movement metrics
1b. Change in EMB trajectories | 3-, 6-, 12-, and 24-months
  Trajectories of investigational EMBs over time
2a. Change in Annual Relapse Rate (ARR) | 12 and 24 months from baseline
  MS relapse is defined as the appearance of a new neurological abnormality or worsening of a previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must have been present for at least 24 hours and must have occurred in the absence of fever (< 37.5°C) or of a known infection.
2b. Change in patient disability measured by Expanded Disability Status Scale EDSS | 3,6,12,24 months from baseline
  The EDSS is an ordinal scale used for assessing neurologic impairment in MS based on a neurological examination. It consists of scores in each of seven functional systems (FSs) and an ambulation score that are then combined to determine the EDSS steps (ranging from 0 [normal] to 10 (death due to MS). The FSs are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral functions
2b. Change in patient disability measured by Timed 25-foot walk test (T25-FW) | 3,6,12,24 months from baseline
  The T25- is an objective quantitative test of neurological function. It is an ambulation measurement assessing speed of walking: a timed (in seconds) walk of 25 feet (7.62 meters)
2b. Change in patient disability measured by the 9-hole peg test (9-HPT) | 3,6,12,24 months from baseline
  The 9- is an objective quantitative test of neurological function. It is measured to assess both right and left arm scores, the metric is the time, in seconds, required to insert and remove nine pegs. The 9-HPT will be administered 4 2 trials per hand, the time for each trial will be averaged with lower times indicating better performance
2c. Change in objective measures of cognitive impairment as measured by the Symbol Digit Modalities Test (SDMT) | 3,6,12,24 months from baseline
  The SDMT is an objective measure of information processing speed and associated cognitive dysfunction in patients with MS. Using a reference key, the patient has 90 seconds to pair specific numbers with given geometric figures in writing. The raw score corresponds to the total number of correct substitutions, ranging between 0 and 110 with higher scores indicative of better performance.
2c. Change in objective measures of cognitive impairment as measured by the Brief Visuospatial Memory Test (BVMT-R) | 3,6,12,24 months from baseline
  The BVMT-R is a measure of visuospatial learning, the test consists of six abstract symbols on a sheet of paper. Participants are given ten seconds to study the figures and then try to draw them in the same order on a blank page. Performance is scored on accuracy and location with 0-2 points per symbol for a maximum of 12 points per trial. Patients are asked to repeat the task three times with higher scores indicative of better performance
2c. Change in objective measures of cognitive impairment as measured by the Rey Auditory Verbal Learning Test (RAVLT) | 3,6,12,24 months from baseline
  The RAVLT is a test of verbal memory that requires the participant to learn and recall a list of 15 words that are orally presented. This test measures learning across five trials, retrieval of the target list after presenting a distracter list and a 30-minute delay, followed by recognition of the target words from among distracter words such as semantic and phonemic foils. The total learning score is the sum of correct answers across the five trials, with higher scores indicative of better performance.
3a. Association between EMB and annual relapse rate (AAR) | 12 and 24 months
  Association of change in each investigational EMB and ARR established at 12 and 24. To estimate the association of change between each investigational EMB and ARR a Poisson or Negative Binomial Generalized Linear Mixed Model (GLMM) will be used. The metric to assess the association of change over time between each investigational EMB and the outcome variable will be the fixed effect of investigational EMB on ARR, as estimated by the GLMM
3b. Association of EMBs and objective measures of disability - EDSS, T25-FW, and 9-HPT | Up to 24 months
  Longitudinal associations of EMBs and objective measures of disability as measured by the EDSS, T25-FW, and 9-HPT. To estimate the longitudinal associations of change between investigational EMBs and measures of disability as measured by EDSS, T25-FW, and 9-HPT scores Linear Mixed Models (LMMs) with a random intercept will be used. The metric to assess the association of change over time between each investigational EMB and the outcome variable will be the population average fixed effect of each investigational EMB on the outcome, as estimated by the corresponding LMM
3c. Association of EMBs and objective measures of cognitive impairment - SDMT | Up to 24 months
  Longitudinal associations of EMBs and objective measures of cognitive impairment as measured by the SDMT. To estimate the longitudinal associations of change between investigational EMBs and SDMT scores, Poisson GLMMs with a log link and a random intercept will be used. The metric to assess the association of change over time of investigational EMBs and the outcome variables will be the fixed effect of investigational EMBs on the outcomes, as estimated by the GLMMs
3c. Association of EMBs and objective measures of cognitive impairment - BVMT-R, and RAVLT | Up to 24 months
  Longitudinal associations of EMBs and objective measures of cognitive impairment as measured by the BVMT-R and RAVLT. To estimate the longitudinal associations of change between investigational EMBs and measures of disability as measured by EDSS, T25-FW, and 9-HPT scores Linear Mixed Models (LMMs) with a random intercept will be used. The metric to assess the association of change over time between each investigational EMB and the outcome variable will be the population average fixed effect of each investigational EMB on the outcome, as estimated by the corresponding LMM
4. Change in serum Neurofilament light Chain (sNfL) | 3,6,12,24 months from baseline
  Change in NfL concentration in serum
5a. Change in patient-reported physical and psychological impact of MS disease as measured by the Multiple Sclerosis impact scale-29 version 2 (MSIS-29v2) | 3,6,12,24 months from baseline
  The MSIS-29v2 is a PRO measure that evaluates the physical and psychological effects of living with MS. The questionnaire consists of 29 items and is scored from 0 to 100, with higher scores indicating a more significant impact of MS.
  The measure is divided into two subscales: a physical impact scale of 20 items, and a psychological impact scale of 9 items. All items consist of a four-point Likert-type response format: "not at all;" "a little;" "moderately;" and "extremely."
5b. Baseline assessment and change in patient-reported depression as measured by the Beck depression inventory-II (BDI-II) | 3,6,12,24 months from baseline
  The BDI-II scale is a measure that evaluates depression in patients with MS. It is a self-reported questionnaire that consists of 21 items that measures characteristic attitudes and symptoms of depression. Each item is scored 0 to 3 points for a total score range of 0 to 63. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression
5c. Change in patient-reported cognitive impairment as measured by the MS neuropsychology questionnaire (MSNQ) | 3,6,12,24 months from baseline
  The MSNQ is a PRO that assesses perceived cognitive impairment among people with MS. It consists of 15 questions that cover different aspects of cognitive function, such as attention, planning, and language. The questions use a scale from 0 (never) to 4 (frequently) to indicate the frequency of cognitive difficulties.
5d. Change in patient-reported mobility as measured by the MS walking scale-12 version 1 (MSWS-12v1) | 3,6,12,24 months from baseline
  The 12-item MSWS is a PRO measure of the impact of MS on walking ability. The MSWS-12 consists of 12 questions that assess how much MS affects various aspects of walking, such as speed, balance, distance, and effort. The MSWS-12 is scored on a scale from 0 to 100, with higher scores indicating greater impairment
6. Incidence of treatment emergent adverse events and serious adverse events | 24 months
  Percentage of participants reporting treatment emergent adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Novartis Pharmaceuticals
Locations (8):
- Canada (8):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Sydney, Nova Scotia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com